CLINICAL TRIAL: NCT05209165
Title: Semaglutide as Treatment of Overweight and Obese Individuals to Reduce Atrial Fibrillation Burden
Brief Title: Semaglutide to Reduce Atrial Fibrillation Burden
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Company decision
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adam Oesterle, Principal Investigator, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFVAEP1
Record Dates: First submitted 2022-01-14; First posted 2022-01-26 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Obesity; Overweight
Keywords: weight loss; atrial fibrillation; lifestyle modification
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Overweight; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — weekly Semaglutide (increased from starting dose of 0.25 mg at four-week intervals (0.5 mg, 1.0 mg, 1.7 mg) to a target dose of 2.4 mg) for 52 weeks with intake visit for the VA MOVE program
  Arms: Semaglutide
Drug: Placebo — Matching placebo and intake visit for VA MOVE
  Arms: Placebo

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia worldwide. AF is associated with obesity and the co-morbidities of obesity, including hypertension and obstructive sleep apnea (OSA) which increase left atrial (LA) size and decrease LA function. Semaglutide, a Glucagon-like peptide receptor 1 agonist (GLP-1 RA), is currently approved by the Food and Drug Administration for weight loss for individuals with and without diabetes. The effects of pharmacologic weight loss with Semaglutide on AF are unknown. The investigators plan on conducting a randomized controlled trial of semaglutide versus placebo in individuals with paroxysmal or early persistent AF (>10% AF burden on ambulatory monitoring, a previous electrical cardioversion, or AF lasting ≥ 7 days but < 3 months who have a body mass index ≥ 27.0 kg/m2. The trial will last for 52 weeks. The primary outcome will be the change in AF burden for 2 weeks, immediately before starting the medication or placebo to two weeks starting at week 50, as determined by an implantable loop recorder or two week ambulatory Additional outcomes will be change in epicardial adipose tissue as determined by chest/abdomen/pelvis computed tomography scan at enrollment and at week 52, change in apnea-hypopnea index from baseline sleep study to week 52 sleep study, change in LA longitudinal strain from baseline echocardiogram to echocardiogram at 52 weeks, and change on symptom surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with a BMI ≥ 27 kg/m2 who have paroxysmal AF with a ≥ 10% burden on ambulatory monitoring or a previous electrical cardioversion or early persistent AF (≥ 7 days, < 3 months) who are willing to attempt rhythm control.

Exclusion Criteria:

* Unable to consent
* A personal or family history of medullary thyroid carcinoma
* A personal or family history of multiple endocrine neoplasia syndrome type 2
* History of allergic reaction to Semaglutide or any of its components
* Currently pregnant or planning to become pregnant
* Currently breastfeeding
* History of acute pancreatitis
* History of pancreatic adenocarcinoma
* Previous or current GLP-1 RA use
* Previous or current use of alternative pharmacologic weight loss agents (phentermine, diethylpropion, orlistat, phentermine-topiramate, bupropion- naltrexone, gelesis100, or setmelanotide)
* Unable to tolerate anticoagulation
* History of bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | 52 weeks
  Change in AF burden from the two weeks before starting Semaglutide or placebo to the last two weeks of therapy (starting at week 50). AF burden will be assessed as percent of time in AF for two weeks on an implantable loop recorder. If the patient declines implantable loop recorder placement, an ambulatory 2-week monitor will be used instead.

SECONDARY OUTCOMES:
Epicardial adipose tissue | 52 weeks
  Change in epicardial adipose tissue on non-contrast chest/abdomen CT scans from baseline and week 52
Sleep apnea | 52 weeks
  Change in apnea-hypopnea index from baseline sleep study to sleep study at week 52
Left atrial function | 52 weeks
  The change in LA longitudinal strain from the baseline echocardiogram to the echocardiogram at 52 weeks.
Weight change | 52 weeks
  From baseline to week 52
Adherence and Adverse Events | 52 weeks
  From baseline to week 52
Participation in VA MOVE | 52 weeks
  assess participation
Change in AF burden for four weeks | 52 weeks
  Change in AF burden for 4 weeks before starting the medication to weeks 48-52.
Fat depots | 52 weeks
  change in pericardial, abdominal (visceral and subcutaneous) and hepatic adipose tissue
Left atrial size and function | 52 weeks
  Changes in LA size and function between baseline and week 52 echocardiograms: LA volume as assessed using the biplane disk summation method, LA reservoir strain, LA conduit strain, and LA booster pump strain will be assessed as secondary outcomes
Quality of life on Healthcare Quality of Life surverys | 52 weeks
  Quality of life on the Short-Form 36 survey and the AF symptoms and severity checklist, which will be completed at baseline and at week 52
Change in C-reactive Protein (CRP) | 52 weeks
  Change in the biomarker CRP between baseline and week 52
Blood pressure | 52 weeks
  Changes in blood pressure and blood pressure medication use between baseline and week 52 will be assessed at those visits.
Change in Interleukin-6 (IL-6) | 52 weeks
  Change in the biomarker IL- 6 between baseline and week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Medical Center San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No